CLINICAL TRIAL: NCT07132489
Title: Validation of Novel Metabolic, Inflammatory, and Hepatic-Renal Biomarkers-HbA1c/C-peptide Ratio, Neutrophil/HDL Ratio, and ALBI Score-for Predicting the No-Reflow Phenomenon After Primary PCI in Patients With STEMI.
Brief Title: Validation of New Biomarkers for Predicting No-Reflow in STEMI Patients Undergoing Primary PCI
Acronym: VaBiNoR
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam Eldin Alaa Abdelhafiz mohamed, Principal investigator, cardiology Department, Assiut University
Other Study IDs: New Biomarkers in No-Reflow
Record Dates: First submitted 2025-08-11; First posted 2025-08-20 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Infarction; No Reflow Phenomenon
MeSH Terms: conditions — Myocardial Infarction; No-Reflow Phenomenon

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month

GROUPS / COHORTS (2):
- No-Reflow Group: STEMI patients undergoing primary PCI who develop angiographic no-reflow, defined as final TIMI flow ≤2 and/or Myocardial Blush Grade (MBG) 0-1 after stent deployment in the absence of mechanical obstruction (no dissection, spasm, residual thrombus, or significant residual stenosis). Planned enrollment: 56.
  Interventions: Diagnostic Test: HbA1c/C-peptide ratio Albumin-bilirubin (ALBI) score. Neutrophil/HDL ratio
- Reflow Group: STEMI patients undergoing primary PCI who achieve successful epicardial and microvascular reperfusion, defined as final TIMI 3 flow and MBG 2-3 after PCI. Planned enrollment: 56.
  Interventions: Diagnostic Test: HbA1c/C-peptide ratio Albumin-bilirubin (ALBI) score. Neutrophil/HDL ratio

INTERVENTIONS:
Diagnostic Test: HbA1c/C-peptide ratio Albumin-bilirubin (ALBI) score. Neutrophil/HDL ratio — 1. To investigate whether the HbA1c to C-peptide ratio can serve as a predictive marker for no-reflow, reflecting the impact of chronic glycemic control and pancreatic beta-cell function.
  2. To evaluate the neutrophil-to-HDL ratio as a potential indicator of no-reflow, representing the balance between systemic inflammation and endogenous vascular protection.
  3. To examine the prognostic value of the albumin-bilirubin (ALBI) score in identifying patients at higher risk for no-reflow, considering the systemic influence of hepatic function and inflammation.

SUMMARY:
To evaluate the diagnostic value of the selected emerging biomarkers in predicting the no-reflow phenomenon among patients presenting with STEMI undergoing primary PCI. These biomarkers include:

HbA1c/C-peptide ratio

Albumin-bilirubin (ALBI) score.

Neutrophil/HDL ratio

DETAILED DESCRIPTION:
The no-reflow phenomenon is a well-recognized complication following primary percutaneous coronary intervention (PCI) in patients presenting with ST-segment elevation myocardial infarction (STEMI). Despite successful opening of the occluded coronary artery, impaired myocardial perfusion may persist, significantly increasing the risk of adverse cardiovascular outcomes.

Recent research has identified several novel biomarkers that may help predict the risk of no-reflow. These include metabolic, inflammatory, and hepatic-renal markers that reflect the systemic milieu of patients with acute coronary syndromes. Among these emerging biomarkers, the following are of particular interest:

* HbA1c/C-peptide ratio: Reflects chronic glycemic burden and residual beta-cell function.
* Neutrophil/HDL ratio: A combined marker of inflammation and lipid-associated atheroprotection.
* Albumin-bilirubin (ALBI) score: A composite liver function marker potentially linked to systemic inflammation and perfusion status.

This study aims to validate the prognostic value of these biomarkers in predicting the no-reflow phenomenon in STEMI patients undergoing primary PCI.

To validate the clinical utility of selected emerging biomarkers in predicting the no-reflow phenomenon among patients presenting with ST-segment elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PCI).

Thus , our objective is to investigate :

1. To investigate whether the HbA1c to C-peptide ratio can serve as a predictive marker for no-reflow, reflecting the impact of chronic glycemic control and pancreatic beta-cell function.
2. To evaluate the neutrophil-to-HDL ratio as a potential indicator of no-reflow, representing the balance between systemic inflammation and endogenous vascular protection.
3. To examine the prognostic value of the albumin-bilirubin (ALBI) score in identifying patients at higher risk for no-reflow, considering the systemic influence of hepatic function and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Suitable for and undergoing timely primary PCI based on symptoms and clinical judgment
* Provision of informed consent

Exclusion Criteria:

* History of previous MI, PCI, or CABG
* Known chronic inflammatory or autoimmune diseases
* Advanced renal or hepatic failure
* Active infection or malignancy at presentation
* Incomplete data or refusal to consent

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will include patients presenting with ST-segment elevation myocardial infarction (STEMI) who are admitted to the [specify hospital/center] and undergo primary percutaneous coronary intervention (PCI).
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c/C-peptide ratio predictive accuracy for no-reflow phenomenon | Baseline (prior to PCI)
  Diagnostic accuracy of HbA1c/C-peptide ratio for predicting the no-reflow phenomenon in STEMI patients undergoing primary PCI, assessed by area under the ROC curve (AUC).
Albumin-bilirubin (ALBI) score predictive accuracy for no-reflow phenomenon | Baseline (prior to PCI)
  Diagnostic accuracy of ALBI score for predicting the no-reflow phenomenon in STEMI patients undergoing primary PCI, assessed by area under the ROC curve (AUC).
Neutrophil/HDL ratio predictive accuracy for no-reflow phenomenon | Baseline (prior to PCI)
  Diagnostic accuracy of neutrophil/HDL ratio for predicting the no-reflow phenomenon in STEMI patients undergoing primary PCI, assessed by area under the ROC curve (AUC).

SECONDARY OUTCOMES:
Correlation of HbA1c/C-peptide ratio, Neutrophil-to-HDL ratio, and Albumin-Bilirubin (ALBI) score with in-hospital major adverse cardiovascular events (MACE). | Baseline to hospital discharge.
  HbA1c/C-peptide ratio (unit: ratio, measured from immunoassay-derived HbA1c and C-peptide levels), Neutrophil-to-HDL ratio (unit: ratio, derived from complete blood count and serum HDL measurement), and Albumin-Bilirubin (ALBI) score (unit: score, calculated from serum albumin [g/dL] and total bilirubin [mg/dL]) will be correlated with the incidence of in-hospital major adverse cardiovascular events (MACE) [unit: % of patients experiencing MACE].
Correlation of HbA1c/C-peptide ratio, Neutrophil-to-HDL ratio, and Albumin-Bilirubin (ALBI) score with 1-month major adverse cardiovascular events (MACE). | Baseline to 1-month follow-up.
  HbA1c/C-peptide ratio (unit: ratio, measured from immunoassay-derived HbA1c and C-peptide levels), Neutrophil-to-HDL ratio (unit: ratio, derived from complete blood count and serum HDL measurement), and Albumin-Bilirubin (ALBI) score (unit: score, calculated from serum albumin [g/dL] and total bilirubin [mg/dL]) will be correlated with the incidence of major adverse cardiovascular events (MACE) at 1-month follow-up [unit: % of patients experiencing MACE].

CONTACTS AND LOCATIONS:
Overall Officials: Hossam H. Ali, Principal Investigator